CLINICAL TRIAL: NCT03483077
Title: A Partially Randomised, Single-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Doses of BI 730460 Administered as Tablets to Healthy Subjects, and a Randomised, Open-label, Single-dose, Two-way Cross-over Bioavailability Comparison of BI 730460 as Tablet With and Without Food
Brief Title: This Study in Healthy Volunteers Determines the Amount of BI 730460 in the Blood When Taken as Tablet. It Looks at How Different Doses of BI 730460 Are Taken up in the Body and How Well They Are Tolerated. The Study Also Tests How Food Influences the Amount of BI 730460 in the Blood.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was ended after completion of dose group 6 of the SRD part, in accordance with a predefined protocol discontinuation criteria. The planned bioavailability evaluation was not performed due to the sponsor's decision.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1416-0001; 2017-004446-15 (EudraCT Number)
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Placebo matching BI 730460 (Placebo Comparator): Placebo tablet(s) matching BI 730460 tablet(s) administered orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) - Single rising dose (SRD) part.
  Interventions: Drug: Placebo
- 2 milligram (mg) - BI 730460 (Experimental): A single dose of 2 mg BI 730460 administered as film-coated tablets orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) - Single rising dose (SRD) part.
  Interventions: Drug: BI 730460
- 8 mg - BI 730460 (Experimental): A single dose of 8 mg BI 730460 administered as film-coated tablets orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) - Single rising dose (SRD) part.
  Interventions: Drug: BI 730460
- 25 mg - BI 730460 (Experimental): A single dose of 25 mg BI 730460 administered as film-coated tablets orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) - Single rising dose (SRD) part.
  Interventions: Drug: BI 730460
- 50 mg - BI 730460 (Experimental): A single dose of 50 mg BI 730460 administered as film-coated tablets orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) - Single rising dose (SRD) part.
  Interventions: Drug: BI 730460
- 100 mg - BI 730460 (Experimental): A single dose of 100 mg BI 730460 administered as film-coated tablets orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) - Single rising dose (SRD) part.
  Interventions: Drug: BI 730460
- 200 mg - BI 730460 (Experimental): A single dose of 200 mg BI 730460 administered as film-coated tablets orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) - Single rising dose (SRD) part.
  Interventions: Drug: BI 730460

INTERVENTIONS:
Drug: BI 730460 — tablets
  Arms: 100 mg - BI 730460; 2 milligram (mg) - BI 730460; 200 mg - BI 730460; 25 mg - BI 730460; 50 mg - BI 730460; 8 mg - BI 730460
Drug: Placebo — tablets
  Arms: Placebo matching BI 730460

SUMMARY:
The primary objective of the single-rising dose (SRD) part (trial part 1) is to investigate the safety and tolerability of BI 730460 in healthy subjects following oral administration of single rising doses. The secondary objective is the exploration of the pharmacokinetics (PK) including dose proportionality, and pharmacodynamics of BI 730460 after single dosing.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

- Male subjects with women of childbearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The evaluation of single-rising dose (SRD) of BI 730460 was designed as a partially randomised, single-blind, placebo-controlled trial and the evaluation of bioavailability of BI 730460 with and without food was designed as a randomised, open-label, single-dose, two-way cross-over trial.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo Matching BI 730460 | 2 Milligram (mg) - BI 730460 | 8 mg - BI 730460 | 25 mg - BI 730460 | 50 mg - BI 730460 | 100 mg - BI 730460 | 200 mg - BI 730460
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 12 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: Participants who received at least 1 dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching BI 730460 | 2 Milligram (mg) - BI 730460 | 8 mg - BI 730460 | 25 mg - BI 730460 | 50 mg - BI 730460 | 100 mg - BI 730460 | 200 mg - BI 730460 | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.0 (6.8) | 36.0 (5.3) | 30.3 (6.2) | 30.7 (8.5) | 34.7 (6.7) | 30.5 (4.7) | 33.7 (7.9) | 32.7 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events
Description: Percentages are calculated using total number of participants per treatment as the denominator.
  MedDRA version used for reporting: 22.0.
Time Frame: From drug administration until end of trial, up to 13 days.
Population: Treated set: Participants who received at least 1 dose of trial drug.
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Placebo Matching BI 730460 | 2 Milligram (mg) - BI 730460 | 8 mg - BI 730460 | 25 mg - BI 730460 | 50 mg - BI 730460 | 100 mg - BI 730460 | 200 mg - BI 730460
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Percentage of participants (%) | 8.3 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0 | 0.0

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 730460 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 730460 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: Within 3 hours (h) prior to drug administration followed by 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 24.0, 34.0, 48.0, 72.0, 96.0, 168.0 hours post drug administration.
Population: Pharmacokinetic analysis set: Participants from the treated set receiving BI 730460 who provided at least 1 secondary pharmacokinetic parameter that was not excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomol*hour per litre
Arm/Group | 2 Milligram (mg) - BI 730460 | 8 mg - BI 730460 | 25 mg - BI 730460 | 50 mg - BI 730460 | 100 mg - BI 730460 | 200 mg - BI 730460
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Nanomol*hour per litre | 557 (35.4) | 2540 (41.2) | 5610 (25.4) | 11200 (56.8) | 31500 (23.8) | 47600 (36.1)

3. Secondary Outcome: Maximum Measured Concentration of BI 730460 in Plasma
Description: Maximum measured concentration of BI 730460 in plasma (Cmax).
Time Frame: as for outcome 2
Population: Pharmacokinetic analysis set: Participants from the treated set who received BI 730460 and provided at least 1 secondary pharmacokinetic parameter that was not excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol per litre
Arm/Group | 2 Milligram (mg) - BI 730460 | 8 mg - BI 730460 | 25 mg - BI 730460 | 50 mg - BI 730460 | 100 mg - BI 730460 | 200 mg - BI 730460
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
nanomol per litre | 31.8 (23.2) | 140 (34.0) | 1860 (23.8) | 309 (11.8) | 597 (22.6) | 1470 (32.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from drug administration till end of trial, up to 13 days
Description: Treated Set (TS): Participants who received at least 1 dose of trial drug.
Groups:
- Total on Treatment: Total over all on treatment phases included in this analysis
Arm/Group | Placebo Matching BI 730460 | 2 Milligram (mg) - BI 730460 | 8 mg - BI 730460 | 25 mg - BI 730460 | 50 mg - BI 730460 | 100 mg - BI 730460 | 200 mg - BI 730460 | Total on Treatment
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/48
Other Adverse Events (participants affected / at risk) | 5/12 | 0/6 | 1/6 | 3/6 | 0/6 | 1/6 | 2/6 | 12/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 730460 (N=12) | 2 Milligram (mg) - BI 730460 (N=6) | 8 mg - BI 730460 (N=6) | 25 mg - BI 730460 (N=6) | 50 mg - BI 730460 (N=6) | 100 mg - BI 730460 (N=6) | 200 mg - BI 730460 (N=6) | Total on Treatment (N=48)
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medical device site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
The trial was ended after completion of dose group 6 of the SRD part, in accordance with a predefined protocol discontinuation criteria. The planned bioavailability evaluation was not performed due to the sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT03483077/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT03483077/SAP_001.pdf